CLINICAL TRIAL: NCT04059029
Title: Predictors of Improvement of Nonalcoholic Fatty Liver Disease in Morbidly Obese Patients Undergoing Bariatric Surgery
Brief Title: Nonalcoholic Fatty Liver Disease in Morbidly Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N201601029
Record Dates: First submitted 2016-12-22; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2016-09

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: Nonalcoholic fatty liver disease; morbidly obese; Bariatric surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During bariatric surgery, all patients would undergo a wedge liver biopsy under laparoscopic guidance. The diagnosis of NASH and liver fibrosis would be made histologically. The levels of total cholesterol, low-density lipoprotein, triglyceride, albumin, insulin, glucose, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, C-peptide, iron, calcium, complete blood cell counts would be assessed before and 12 months after bariatric surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morbidly obese patients with NAFLD: Morbidly obese patient with Nonalcoholic fatty liver disease. The starting point for each patient is the day of surgery and the end-point is 1 year after the operation. During bariatric surgery, all patients would undergo a wedge liver biopsy under laparoscopic guidance. The diagnosis of NASH would be made histologically.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — During bariatric surgery, all patients would undergo a wedge liver biopsy under laparoscopic guidance.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of abnormal liver biochemistry tests in the world. The prevalence rate of NAFLD has been reported to be 30-40% in men and 15-20% in women, up to 70% of people with type 2 diabetes mellitus (Type 2 DM) and even surpassing 74% to 90% of morbidly obese patients with body mass index (BMI) higher than 35 kg/m^2. The primary aims of this prospective cohort study would evaluate the predictive factors of successful weight reduction, NAFLD and nonalcoholic steatohepatitis (NASH) improvement in a large cohort of morbidly obese patients undergoing bariatric surgery. Secondarily, the diagnostic accuracy of noninvasive serum markers, doppler ultrasonography and transient elastography would be validated. Thirdly, we would conduct gene expression analyses to elucidate biological pathways underlying NAFLD phenotypes in this unique cohort.

DETAILED DESCRIPTION:
This prospective study have been approved by Taipei Medical University-Joint Institutional Review Board. The starting point for each patient is the day of surgery and the end-point is 1 year after the operation. During bariatric surgery, all patients would undergo a liver biopsy under laparoscopic guidance. The diagnosis of NASH and liver fibrosis would be made histologically. For histological examinations, liver tissue specimens would be fixed in 10 % formalin, embedded in paraffin, and then stained with hematoxylin and eosin. A detailed history wound be obtained including history of alcohol use, type 2 DM, hypertension, or hyperlipidemia. Written informed consents would be obtained from all patients who would agree to undergo surgery. A histologic assessment would be planned approximately 1 year after bariatric surgery, if patient would agree.

In this study, excess weight loss (EWL) is defined as the excess weight over the ideal body weight calculated according to the Metropolitan Life Weight Tables. The weight reduction success would be defined as the percentage of excess weight loss (%EWL) >50% at the point of 1 year after operation. Diagnosis and classification of type 2 DM is based on criteria established by the American Diabetes Association. The individual components of glycemic control (levels of serum glucose, HbA1c levels) body weight, waist circumference, and blood pressure would be examined. Additionally, the levels of total cholesterol, LDL-C, triglyceride, uric acid, aspartate aminotransferase (AST),alanine aminotransferase (ALT), albumin, insulin, C-peptide, iron, calcium, complete blood cell counts would be assessed 1 day before surgery and 12 months post-operatively. All patients would receive abdominal ultrasonography, duplex doppler ultrasonography, transient elastography (FibroScan®) before and 12 months after bariatric surgery. The diagnosis accuracy of transient elastography (FibroScan®) would be validated. Transient elastography (FibroScan®) appears to be a non-invasive, reproducible, and reliable method for predicting liver fibrosis, in patients with hepatitis B virus, hepatitis C virus, NAFLD and alcoholic liver disease.

Patients body weight would be measured in light clothing without shoes to the nearest 0.1 kg, and body height would be measured to the nearest 0.1 cm. BMI is calculated as weight in kilograms divided by height in meters squared. Waist circumference would be measured midway between the lateral lower rib margin and the superior anterior iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female Morbidly obese patients age 20-65 years with BMI over 37.5 kg/m^2, or BMI over 32.5 kg/m^2 with comorbidity other than diabetes (hypertension, NASH, dyslipidemia, obstructive sleep apnea, osteoarthritis joint…etc.) or BMI over 27.5 kg/m^2 with poor control diabetes undergoing bariatric surgery

Exclusion Criteria:

* The presence of end organ damage
* Previous bariatric surgery
* Women who are pregnant or nursing
* Prolonged exposure to known hepatotoxins such as alcohol or drugs
* Concurrent hepatitis B virus, hepatitis C virus, hepatitis D virus, or human immunodeficiency virus infection
* Concurrent autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis
* Wilson disease or hemochromatosis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patient undergoing bariatric surgery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from body mass index (BMI) at 12 months after surgery | pre-surgery and 12 months after surgery
  The BMI would be calculated by dividing the body weight (in kilograms) by the square body height (in meters).

SECONDARY OUTCOMES:
Change from alanine aminotransferase at 12 months after surgery | pre-surgery and 12 months after surgery
  Liver function test
Change from aspartate aminotransferase at 12 months after surgery | pre-surgery and 12 months after surgery
  Liver function test
Nonalcoholic steatohepatitis | 1 day of surgery
  The diagnosis of nonalcoholic steatohepatitis (NASH) would be made histologically. A score for steatosis, activity and fibrosis would be given to each patient for the diagnosis of NASH as in Bedossa's study. (Reference: Hepatology. 2012 Nov;56(5):1751-9.)

CONTACTS AND LOCATIONS:
Overall Officials: Weu Wang, M.D.&PhD, Study Chair — Comprehensive weight management center, Taipei Medical University hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Gastroenterological Association; American Association for the Study of Liver Diseases; American College of Gastroenterologyh. The diagnosis and management of non-alcoholic fatty liver disease: practice guideline by the American Gastroenterological Association, American Association for the Study of Liver Diseases, and American College of Gastroenterology. Gastroenterology. 2012 Jun;142(7):1592-609. doi: 10.1053/j.gastro.2012.04.001. Epub 2012 May 15. No abstract available. PMID 22656328
- [Background] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287
- [Background] Morita S, Neto Dde S, Morita FH, Morita NK, Lobo SM. Prevalence of Non-alcoholic Fatty Liver Disease and Steatohepatitis Risk Factors in Patients Undergoing Bariatric Surgery. Obes Surg. 2015 Dec;25(12):2335-43. doi: 10.1007/s11695-015-1696-5. PMID 25920616
- [Background] Puzziferri N, Roshek TB 3rd, Mayo HG, Gallagher R, Belle SH, Livingston EH. Long-term follow-up after bariatric surgery: a systematic review. JAMA. 2014 Sep 3;312(9):934-42. doi: 10.1001/jama.2014.10706. PMID 25182102
- [Background] Arterburn D, Powers JD, Toh S, Polsky S, Butler MG, Portz JD, Donahoo WT, Herrinton L, Williams RJ, Vijayadeva V, Fisher D, Bayliss EA. Comparative effectiveness of laparoscopic adjustable gastric banding vs laparoscopic gastric bypass. JAMA Surg. 2014 Dec;149(12):1279-87. doi: 10.1001/jamasurg.2014.1674. PMID 25353723
- [Background] Lee WJ, Almulaifi A, Chong K, Chen SC, Tsou JJ, Ser KH, Lee YC, Chen JC. The Effect and Predictive Score of Gastric Bypass and Sleeve Gastrectomy on Type 2 Diabetes Mellitus Patients with BMI < 30 kg/m(2). Obes Surg. 2015 Oct;25(10):1772-8. doi: 10.1007/s11695-015-1603-0. PMID 25676157
- [Derived] Kao WY, Lin YF, Chang IW, Chen CL, Tang JH, Chang CC, Chang YJ, Wang W. Interleukin-2 receptor alpha as a biomarker for nonalcoholic fatty liver disease diagnosis. J Chin Med Assoc. 2021 Mar 1;84(3):261-266. doi: 10.1097/JCMA.0000000000000469. PMID 33306598